CLINICAL TRIAL: NCT05446233
Title: Single Dose Absorption, Distribution, Metabolism, and Excretion Study of [14C] Antaitavir Hasophate in Healthy Male Participants
Brief Title: ADME Study of [14C] Antaitavir Hasophate in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HEC74647-P-04/CRC-C2222
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-11

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] Antaitavir Hasophate (Experimental): Eligible healthy male subjects received a single oral 100 mg (radioactivity of 200µCi) dose of [14C] Antaitavir Hasophate
  Interventions: Drug: [14C] Antaitavir Hasophate

INTERVENTIONS:
Drug: [14C] Antaitavir Hasophate — 100 mg suspension containing 200µCi of [14C] Antaitavir Hasophate

SUMMARY:
This is a single-centre, open-label, mass balance and biotransformation study in healthy male subjects utilising a single oral dose of [14C] Antaitavir Hasophate.

ELIGIBILITY:
Inclusion Criteria:

* signing of informed consent
* Weight: Body mass index (BMI) is 19.0~28.0 kg/m2
* Subjects are able to communicate well with the investigators and be able to complete the trial according to the process

Exclusion Criteria:

* Those who are known to have allergy history or allergy constitution to the test preparation and any of its components or related preparations
* Positive test for hepatitis B (surface antigens HBs), or C (antibody HCs), positive test for HIV, Treponema pallidum antibody positive
* Positive results from urine drug screen test
* Donate blood or lose blood 400 mL or more within 3 month prior to dosing
* Subjects who have used any medication, biological product, Chinese patent medicine, herbal medicine, nutritional supplements or health care products within 14 days prior to the first dose of study medication, or participated in other clinical studies or participated in a clinical study of test preparation within 3 months prior to the first dose of study medication
* History of needles or blood fainting, or have difficulty in blood collection or cannot tolerate venipuncture for blood collection

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Distribution ratio of total radioactivity in whole blood and plasma of [14C] Antaitavir Hasophate | up to 15 days
  To investigate the pharmacokinetics of total radioactivity in plasma after oral [14C] Antaitavir Hasophate in healthy subjects, and the distribution ratio of total radioactivity in whole blood and plasma
Cumulative excretion of [14C] Antaitavir Hasophate -related material (radioactivity in plasma, urine and fecal samples) | up to 15 days
  Percent (%) of each radiolabeled drug-related material (parent and each metabolite) will be determined in plasma, urine and feces.

SECONDARY OUTCOMES:
Identification of the Proportion of different metabolites to determine biotransformation pathway of Antaitavir Hasophate | up to 15 days
  Proportion of different metabolites(Antaitavir Hasophate and main metabolites）
Quantitive analysis of the concentrations of Antaitavir Hasophate and main metabolites in plasma using the validated LC-MS/MS to obtain pharmacokinetic data | up to 15 days
  The concentrations of Antaitavir Hasophate and main metabolites in plasma
Number of adverse events (AE) experienced by subjects | up to 15 days
  To examine the safety and tolerability of [14C] Antaitavir Hasophate given orally

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai xuhui central hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No